CLINICAL TRIAL: NCT04585035
Title: A Phase 1/2, Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of D-1553 in Subjects With Advanced or Metastatic Solid Tumors With KRasG12C Mutation
Brief Title: Study to Evaluate D-1553 in Subjects With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D1553-101; KEYNOTE-C15 MK3475-C15 (Other: Merck Sharpe and Dohme LLC)
Record Dates: First submitted 2020-09-27; First posted 2020-10-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor, Adult; NSCLC; CRC
MeSH Terms: interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Intervention Model Description: Phase Ia dose escalation portion of the study followed by a Phase Ib dose combination portion. Phase 2 will consist of 5 treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation of D-1553 monotherapy (Experimental): Phase 1a will evaluate up to 7 sequential cohorts with different doses of D-1553 to determine safety, tolerability, MTD and RDE in patients with solid tumors with KRasG12C mutation.
  Interventions: Drug: D-1553
- Dose combination of D-1553 with other therapies (Experimental): Phase 1b will determine the MTD of D-1553 in combination treatment in subjects with advanced or metastatic NSCLC, CRC and other solid tumors. There are multiple groups in Phase 1b for different tumor types and treatment combinations to evaluate safety, MTD and RP2D.
  Interventions: Drug: D-1553; Drug: D-1553 in combination with Drug: pembrolizumab, Drug:KEYTRUDA® , Drug: cetuximab, Drug: other
- Phase 2 of D-1553 monotherapy and combination therapies (Experimental): The Phase 2 portion is a multi-arm, parallel, open label study to evaluate the efficacy of D- 1553 single agent and combination treatments in subjects with advanced or metastatic solid tumors with KRas G12C mutation. Enrollment into phase 2 will be opened after confirmation of the recommended phase 2 dose.
  Interventions: Drug: D-1553; Drug: D-1553 in combination with Drug: pembrolizumab, Drug:KEYTRUDA® , Drug: cetuximab, Drug: other

INTERVENTIONS:
Drug: D-1553 — D-1553 is a novel, targeted KRasG12C inhibitor that is being developed as a potential oral agent for advanced or metastatic solid tumors with KRasG12C mutation.
Drug: D-1553 in combination with Drug: pembrolizumab, Drug:KEYTRUDA® , Drug: cetuximab, Drug: other — Standard treatment of solid tumor, NSCLC or CRC
  Arms: Dose combination of D-1553 with other therapies; Phase 2 of D-1553 monotherapy and combination therapies

SUMMARY:
This is a phase 1/2, open label study of D-1553 single agent and combination treatment to assess the safety and tolerability, identify the MTD and RP2D, evaluate the PK properties and antitumor activities in subjects with advanced or metastatic solid tumor with KRasG12C mutation.

ELIGIBILITY:
Inclusion criteria

* Subject with histologically proven, locally advanced, unresectable and/or metastatic solid tumor, for which no standard treatment is available, or the subject is refractory to or intolerant of existing standard treatment.
* Subject has KRasG12C mutation in tumor tissue or other bio-specimens containing cancer cells or DNA. Historical, local laboratory result (up to 5 years prior to this study) can be used for Phase 1 subjects. Phase 2 subjects must be tested for KRasG12C mutation by a central laboratory.
* Subject has tumor type requirement as follows: advanced or metastatic solid tumors including NSCLC and CRC.
* Subject has measurable disease according to RECIST, v1.1.

Exclusion Criteria:

* Subject with unstable or progressive central nervous system (CNS) metastases.
* Subject with acute myocardial infarction, severe/unstable angina; or with cardiac insufficiency of New York Heart Association Functional Classification Grade 2 or above.
* Subject has corrected QT interval using Fridericia's formula (QTcF) prolongation at rest, where the mean QTc interval is > 480 msec based on triplicate measurements of electrocardiogram (ECG).
* Subject with stroke or other severe cerebrovascular diseases within 12 months before enrollment;
* Subject with interstitial lung disease or acute lung infection not yet recovered including but not limited to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection;
* Subject has any history or evidence of substance abuse or medical, psychological or social conditions that may, in the opinion of the investigator, interfere with participation in the study or evaluation of the study results.
* Subject has impaired gastrointestinal (GI) function or GI diseases that may significantly alter the absorption or metabolism of oral medications.
* Subject has unresolved toxicities from prior anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI CTCAE, v5.0, Grade ≤ 1 (Grade ≤ 2 for peripheral neuropathy).
* Subject had major surgery within 4 weeks prior to study intervention administration or last dose of palliative radiation therapy within 2 weeks prior to study intervention administration.
* Subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subject incidence of Dose-limiting toxicities (DLT) | through out the DLT period, approximately 21 days
Number of subjects participants with adverse events | Through study completion, approximately 3 years
Plasma concentration of D-1553 as a single agent or in combination with other therapies in subjects wiht advanced or metastatic solid tumors with KRas G12C mutation. | Through study completion, approximately 3 years

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - Research Site, Fresno, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Louisville, Kentucky
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
- Australia (9):
  - Research Site, Blacktown, New South Wales
  - Research Site, East Albury, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Waratah, New South Wales
  - Research Site, Woodville South, South Australia
  - Research Site, Fitzroy, Victoria
  - Research Site, Frankston, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Nedlands, Western Australia
- South Korea (3):
  - Research Site, Seogu, Busan
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Seoul
- Taiwan (3):
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan DY, Wu HX, Xu Y, Munster PN, Deng Y, Richardson G, Yan D, Lee MA, Lee KW, Pan H, Hager S, Li X, Wei S, Hou X, Underhill C, Millward M, Nordman I, Zhang J, Shan J, Han G, Grewal J, Gadgeel SM, Sanborn RE, Huh SJ, Hu X, Zhang Y, Xiang Z, Luo L, Xie X, Shi Z, Wang Y, Zhang L, Wang F, Xu RH. Garsorasib, a KRAS G12C inhibitor, with or without cetuximab, an EGFR antibody, in colorectal cancer cohorts of a phase II trial in advanced solid tumors with KRAS G12C mutation. Signal Transduct Target Ther. 2025 Jun 17;10(1):189. doi: 10.1038/s41392-025-02274-z. PMID 40523897